CLINICAL TRIAL: NCT01954758
Title: Clinical Study, International, Multicentre, Prospective, Randomised, Interventional and Controlled, Comparing Fresh Embryo Transfer (ET) Versus Frozen Embryo Transfer (FET) and Personalised Embryo Transfer (pET) Guided by the ERA (Endometrial Receptivity Analysis) Test as a Diagnostic Tool in Patients Treated by IVF/ICSI (in Vitro Fertilisation; Intra-cytoplasmic Sperm Injection)
Brief Title: The ERA Test as a Diagnostic Guide for Personalized Embryo Transfer
Acronym: ERA RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Scientific Director IGENOMIX; Gynaecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1304-C-107-CS
Record Dates: First submitted 2013-09-26; First posted 2013-10-07 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Endometrial Receptivity
Keywords: Window of implantation; Personalized embryo transfer; Fresh embryo transfer; Delayed embryo transfer; Elective deferred embryo transfer; Endometrial receptivity array; Endometrial receptivity analysis; Endometrial receptivity test; Frozen embryo transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized embryo transfer (pET) (Experimental): Patients will undergo a cycle of endometrial preparation following hormone replacement therapy (HRT) and an endometrial biopsy in a substituted cycle after 5 days (around 120 hours) of progesterone administration. The ERA test will determine the window of implantation (WOI) for each patient and will recommend the best time for embryo transfer thereby increasing the chances of a successful outcome. In some specific cases (≤ 10%) a second biopsy will be required to help the bioinformatic predictor to ensure the most appropriated moment for the embryo transfer. In a different cycle, patients will undergo a cycle of controlled ovarian stimulation (COS) to obtain oocytes which will be fertilized by IVF/ICSI and vitrified. In a subsequent cycle, following the ERA result, a personalized embryo transfer (pET) will be carried out following the same conditions in which the ERA test was obtained, using 1 or 2 viable blastocysts previously obtained (day 5 or 6 stage)
  Interventions: Other: personalized Embryo Transfer (pET)
- Frozen embryo transfer (FET) (Active Comparator): Patients will undergo a cycle of controlled ovarian stimulation (COS) to obtain oocytes which will be fertilized by IVF/ICSI. In a subsequent cycle, following hormone replacement therapy (HRT), a frozen embryo transfer (FET) will be performed using 1 or 2 viable blastocysts previously obtained (day 5 or 6 stage).
  Interventions: Other: Frozen Embryo Transfer (FET)
- Fresh embryo transfer (ET) (Active Comparator): Patients will undergo a controlled ovarian stimulation cycle (COS) to obtain oocytes which will be fertilized by IVF/ICSI. In the same cycle, a fresh embryo transfer will be performed using 1 or 2 viable blastocysts previously obtained (day 5 or 6 stage).
  Interventions: Other: Fresh Embryo Transfer (ET)

INTERVENTIONS:
Other: personalized Embryo Transfer (pET)
  Arms: Personalized embryo transfer (pET)
Other: Frozen Embryo Transfer (FET)
  Arms: Frozen embryo transfer (FET)
Other: Fresh Embryo Transfer (ET)
  Arms: Fresh embryo transfer (ET)

SUMMARY:
This project seeks to demonstrate the clinical value of the personalised diagnosis of the endometrial factor in infertility.

DETAILED DESCRIPTION:
This project seeks to investigate differences in implantation (IR), pregnancy (PR), ongoing pregnancy (OP) rates, miscarriages, deliveries (LB) and obstetrical, delivery and neonatal outcomes among women undergoing IVF treatment with own oocytes, at first site appointment (up to 3 previous implantation failures in other sites) and blastocyst stage (day 5 or 6). Patients are allocated through computer-generated randomization into one of the three groups: Fresh embryo transfer (ET), Frozen embryo transfer (FET) or personalized embryo transfer (pET) after identification of the personalized window of implantation using the endometrial receptivity analysis (ERA) test, all of them following the usual clinical practice in a same-cycle embryo transfer.

A total of 546 infertile women under 38 years old undergoing her first IVF/ICSI cycle with elective blastocyst transfer are randomized in this prospective, multicenter, open label and controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients indicated to undergo a cycle of IVF/ICSI with their own oocytes.
2. Age ≤ 37 years
3. BMI: 18.5 to 30
4. Normal ovarian reserve (AFC ≥ 8; FSH < 8)
5. The most appropriated stimulation protocol will be decided by their doctor.
6. Blastocyst transfer (on day 5 or 6)
7. Blastocyst vitrification with open protocols (Cryotop, Cryoleaf, or Cryolock) or closed protocols (Cryotip or CBSStraw.)
8. Any pathology affecting the endometrial cavity such as polyps/sub-mucosal myomas, intramural myomas > 4 cm, or hydrosalpinx affecting the endometrial cavity must be previously operated.

Exclusion Criteria:

1. Patients with recurrent miscarriages (> 2 previous biochemical pregnancies or > 2 spontaneous miscarriages)
2. Patients with a severe male factor (spermatozoa < 2 million/ml)
3. Patients with implantation failure (>3 failed cycles with good quality embryos)

Post-Randomization Exclusion Criteria:

1. Endogenous progesterone level ≥ 1,5 ng/ml at the day of hCG administration in all groups.
2. Absence of blastocysts (day 5 or 6) for embryo transfer.
3. Risk of ovarian hyperstimulation syndrome in any of the three groups and therefore a clinical indication to cancel the transfer cycle where the stimulated patient is from group A (ET).

Note: PGT-A is not an inclusion criteria neither an exclusion criteria, therefore those cycles in which PGT-A was performed will be included

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing IVF treatment
Enrollment: 569 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Live birth delivery rate | 40 weeks
  Percentage of deliveries that resulted in at least one live birth per embryo transfer.

SECONDARY OUTCOMES:
Implantation rate | 12 weeks
  The percentage of gestational sacs observed divided by the number of embryos transferred
Pregnancy rate | 20 weeks
  The percentage of positive pregnancy test divided by the number of embryo transfers
Biochemical pregnancies | 20 weeks
  A pregnancy diagnosed only by the detection of beta hCG in serum
Ectopic pregnancies | 20 weeks
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology
Clinical miscarriages | 20 weeks
  Spontaneous loss of a clinical pregnancy before 20 completed weeks of gestational age
Cumulative pregnancy rate | 12 months
  Cumulative pregnancy rate in the 12 months after the first study embryo transfer
Cumulative implantation rate | 12 months
  Cumulative implantation rate in the 12 months after the first study embryo transfer
Cumulative live birth delivery rate | 12 months
  Cumulative live birth delivery rate per embryo transfer in the 12 months after the first study embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MDPhD, Principal Investigator — IVI Valencia / Igenomix
Locations (16):
- Centre of Reproductive Medicine UZ Brussles, Brussels, Belgium
- Brazil (3):
  - Centro de Infertilidade e Medicina Fetal do Norte Fluminence, Campos dos Goytacazes, Rio de Janeiro
  - Centro de Reproduçao Humana Nilo Frantz, Porto Alegre, Rio Grande do Sul
  - Centro de Reprodução Governador Mario Covas, São Paulo
- Sofia Hospital of Reproductive Medicine - SBALAGRM, Sofia, Bulgaria
- Oak Clinic Sumiyoshi, Osaka, Japan
- IVI Panama, Panama City, Panama
- Spain (8):
  - IVI Bilbao, Leioa, Bizkaia
  - IVI Madrid, Aravaca, Madrid
  - IVI Vigo, Vigo, Pontevedra
  - IVI Alicante, Alicante
  - IVI Barcelona, Barcelona
  - ProcreaTec, Madrid
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia
- Bahceci Health Group, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Katzorke N, Vilella F, Ruiz M, Krussel JS, Simon C. Diagnosis of Endometrial-Factor Infertility: Current Approaches and New Avenues for Research. Geburtshilfe Frauenheilkd. 2016 Jun;76(6):699-703. doi: 10.1055/s-0042-103752. PMID 27365540